CLINICAL TRIAL: NCT03582826
Title: Dynamics of the Gut Microbiota in Idiopathic Malodor Production
Brief Title: Microbial Basis of Systemic Malodor and "People Allergic To Me" Conditions
Acronym: PATM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mebo Research, Inc. (Other)
Collaborators: uBiome (Industry); Aurametrix (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 201805110018MEBO
Record Dates: First submitted 2018-06-11; First posted 2018-07-11 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Nutritional and Metabolic Diseases
Keywords: systemic malodor; body odor; bad breath; PATM; microbiome; TMAU; Malabsorption; Dysbiosis
MeSH Terms: conditions — Nutritional and Metabolic Diseases; Body Odor; Halitosis; Malabsorption Syndromes; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEBO/PATM cohort (Experimental): Nutrition counselling and stress-management counselling behavioral interventions will be given to minimize subjects symptoms and observe corresponding changes in their microbiomes.
  The following subcohorts were formed for analyses of different outcomes: MEBO and PATM subcohorts, TMAU positive and negative subcohorts, Active MEBO, Active PATM, Regression and Remission; MEBO/PATM Cohort that Submitted Gut Samples, MEBO/PATM cohort that answered QoL survey, MEBO/PATM Subcohort that observed and documented both flareups and improvements.
  Interventions: Behavioral: Nutritional counselling; Behavioral: Stress-reduction counseling
- non-MEBO cohort (No Intervention): Data volunteers that never experienced episodes of uncontrollable socially debilitating metabolic body odor (MEBO) or PATM

INTERVENTIONS:
Behavioral: Nutritional counselling — Behavioral nutritional counselling delivered via the Internet.
  Arms: MEBO/PATM cohort
Behavioral: Stress-reduction counseling — The psycho-behavioral intervention includes administering questionnaires and monthly maintenance psychological support delivered via the Internet.
  Arms: MEBO/PATM cohort

SUMMARY:
The purpose of this study is to identify microbial signatures associated with remission and recurrence of idiopathic malodor and PATM conditions.

DETAILED DESCRIPTION:
Human odorprints, mostly owing to the microbiome, have proven their value as biomarkers of health and environmental exposures. In recent years, microbial networks responsible for localized malodors such as halitosis or axillary odor have been mapped by using next generation sequencing approaches. Intestinal microbes responsible for psychologically debilitating systemic malodor (whole-body and extraoral halitosis), however, remain to be identified. Even a relatively straightforward disorder of choline metabolism trimethylaminuria (TMAU) is thought to exhibit complex host-gene microbiome interactions and has not been sufficiently studied.

Proposed controlled pilot study aims to explore the dynamics of microbial communities in remission and flare-up periods. Better knowledge of the important aspects of disease fluctuation should enhance patient care and, combined with our prior data, will help to develop new therapies and treatments.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic malodor or PATM symptoms experienced over a period of several months or years
* able to read and understand the study information
* willing and able to comply with questionnaires, nutritional recommendations, and other study procedures

Exclusion Criteria:

* consistent inability to communicate and process things related to their symptoms
* consistent inability to distinguish physical symptoms from pure emotional reactions
* lack of motivation to start feeling better

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-06-16 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Gabashvili, PhD, Principal Investigator — MeBO Research
Locations (2):
- MeBO Research, Miami, Florida, United States
- MeBO Research LTD, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified patient data will be made partially available when approved by the study sponsor.
Supporting Information: Study Protocol, ICF
Time Frame: one year after completion of the study
Access Criteria: undecided

REFERENCES:
- [Result] Gabashvili IS Cutaneous Bacteria in the Gut Microbiome as Biomarkers of Systemic Malodor and People Are Allergic to Me (PATM) Conditions: Insights From a Virtually Conducted Clinical Trial JMIR Dermatol 2020;3(1):e10508 URL: http://derma.jmir.org/2020/1/e10508/ doi: 10.2196/10508
- See also: uBiome Awards Grant to MEBO Research — https://www.prweb.com/releases/ubiome_awards_grant_to_mebo_research_a_public_charity_to_study_the_dynamic_of_gut_microbiota_in_idiopathic_malodor_production/prweb15949159.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- MEBO/PATM Cohort: The cohort is individuals who experienced symptoms of idiopathic malodor (MEBO) and/or PATM ("people allergic to me" condition)
- Non-MEBO/PATM Cohort: Individuals that never experienced MEBO or PATM symptoms that donated their gut microbiome samples
Period: Overall Study
Arm/Group | MEBO/PATM Cohort | Non-MEBO/PATM Cohort
Started | 119 | 6
Completed (submitted stool samples) | 78 | 6
Not Completed | 41 | 0
Not completed — Lost to Follow-up | 39 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants at Baseline who consented to submit their data
Groups:
- MEBO/PATM Cohort: The cohort is 119 individuals who experienced symptoms of idiopathic malodor (MEBO: 70 participants) and/or PATM ("people allergic to me" condition: 39 participants)
- Non-MEBO/PATM Cohort: 6 data volunteers that never experienced episodes of uncontrollable socially debilitating odor or PATM.
- Total: Total of all reporting groups
Arm/Group | MEBO/PATM Cohort | Non-MEBO/PATM Cohort | Total
Number analyzed (Participants) | 119 | 6 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12) | 40 (20) | 40 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 1 | 80
  Male | 40 | 5 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Number of participants at Baseline who consented to submit their data
  participants
    United States | 70 | 5 | 75
    United Kingdom | 10 | 0 | 10
    Argentina | 4 | 0 | 4
    Brazil | 4 | 0 | 4
    Burkina Faso | 1 | 0 | 1
    Canada | 5 | 0 | 5
    Colombia | 1 | 0 | 1
    France | 1 | 0 | 1
    Hong Kong | 2 | 0 | 2
    Italy | 1 | 0 | 1
    Kenya | 2 | 0 | 2
    Mexico | 1 | 0 | 1
    Morocco | 1 | 0 | 1
    Netherlands | 1 | 0 | 1
    Nigeria | 3 | 0 | 3
    Pakistan | 1 | 0 | 1
    Peru | 2 | 0 | 2
    Philippines | 1 | 0 | 1
    Portugal | 1 | 0 | 1
    South Africa | 1 | 0 | 1
    Spain | 5 | 1 | 6
    Sweden | 1 | 0 | 1
TMAU status [Count of Participants; unit: Participants] — Trimethylaminuria diagnosis at baseline, based on laboratory testing
  Participants
    Primary TMAU | 23 | 0 | 23
    Secondary TMAU | 12 | 0 | 12
    Negative TMAU test result | 26 | 0 | 26
    Not tested for TMAU | 58 | 6 | 64
PATM status [Count of Participants; unit: Participants] — Self-diagnosis of "Metabolic Body Odor" (MEBO) and "People are Allergic to me" (PATM) conditions at baseline
  Participants
    PATM with or without MEBO | 60 | 0 | 60
    MEBO | 59 | 0 | 59
    neither MEBO nor PATM | 0 | 6 | 6

OUTCOME MEASURES:

1. Primary Outcome: Gut Microbiome
Description: Abundance [operational taxonomic units]
Time Frame: 1 year
Population: Study volunteers that submitted gut microbiome samples (84 out of 125 enrolled)
Measure: Mean (95% Confidence Interval); unit: Normalized OTU counts
Units Other Than Participants: samples
Groups:
- MEBO/PATM Cohort That Submitted Gut Samples: Participants who had experienced uncontrollable socially debilitating odor or PATM symptoms and submitted at least one gut sample for analysis (78 out of 119 in MEBO/PATM cohort)
- Non-MEBO/PATM Cohort: Samples of volunteers that never experienced episodes of uncontrollable socially debilitating odor or PATM.
Arm/Group | MEBO/PATM Cohort That Submitted Gut Samples | Non-MEBO/PATM Cohort
Number analyzed (Participants) | 78 | 6
Number analyzed (samples) | 217 | 16
Normalized OTU counts
  Phylum Firmicutes | 52 [50 to 53] | 64 [63 to 65]
  Phylum Bacteroidetes | 25 [24 to 26] | 33 [32 to 34]
  Phylum Tenericutes | 0.04 [0.01 to 0.07] | 0.35 [0.26 to 0.42]
  Phylum Actinobacteria | 3.73 [3.25 to 4.22] | 3.37 [3.06 to 3.67]
  Phylum Proteobacteria | 4.64 [4.07 to 5.22] | 3.70 [3.21 to 4.18]

2. Secondary Outcome: Quality of Life [Score]
Description: QoL: Scores range from 20 (lowest level of satisfaction with life) to 150 (maximal life satisfaction). Quality of life (QOL) will be measured with MEBO quality of life assessment questionnaire, a new tool designed on the basis of the Halitosis Associated Life-quality Test (HALT), Dermatology Life Quality Index (DLQI) and WHOQOL-100 questionnaires. Most questions were devised with a Likert scale of 0-5 where a higher score indicated a higher quality of life. Scores for five negatively framed questions are transformed to positively framed questions. Total QOL score (minimum score of 20 and maximum score of 150) is computed based on four aspects of QOL: physical health, psychological health, social support and environment.
Time Frame: 1 year
Population: Study participants from MEBO/PATM cohort that answered QoL survey (71 out of 119 in MEBO/PATM cohort). Since QOL questionnaire was administered multiple times for each participant, type of units analyzed is number of QoL submissions. Non MEBO/PATM cohort did not participate in this intervention.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: QoL entries
Groups:
- Subjects With Active MEBO/PATM: Individuals experiencing uncontrollable episodes of MEBO or PATM who submitted responses to Quality of Life (QoL) questionnaire.
- Subjects in Regression or Remission: Individuals self-describing themselves as being in remission or regression of MEBO/PATM (experiencing fewer and less severe flareups or disappearance of the symptoms) who submitted responses to QoL questionnaire.
Arm/Group | Subjects With Active MEBO/PATM | Subjects in Regression or Remission
Number analyzed (Participants) | 64 | 7
Number analyzed (QoL entries) | 154 | 34
score on a scale | 57 [55 to 59] | 97 [90 to 105]

3. Secondary Outcome: Idiopathic Malodor Episodes
Description: The number of flareups after study enrollment
Time Frame: 1 year after study enrollment
Population: Individuals from MEBO/PATM cohort who submitted at least one gut microbiome sample accompanied by a QoL survey. Non-MEBO Cohort is not included since they never experienced MEBO/PATM flareups.
Measure: Count of Units; unit: observations
Units Other Than Participants: observations
Groups:
- Subjects With Active MEBO/PATM: Observations of individuals experiencing uncontrollable episodes of malodor or PATM
- Subjects in Regression or Remission: Observations of individuals self-reporting remission or regression of MEBO/PATM (lessening of the severity or disappearance of the symptoms)
Arm/Group | Subjects With Active MEBO/PATM | Subjects in Regression or Remission
Number analyzed (Participants) | 64 | 7
Number analyzed (observations) | 154 | 34
observations
  severe flareups | 81 | 7
  moderate flareups | 27 | 12
  remission episodes | 6 | 12
  not sure | 40 | 3

4. Secondary Outcome: Change in Fecal Microbiome Composition Between Flare-ups and Improvements
Description: The fecal microbial composition will be measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing of submitted gut samples
Time Frame: 1 year
Population: Study participants that submitted two or more microbiome samples (each accompanied by answers to QoL questionnaire) and observed improvement of their symptoms (22 participants that documented their improvement out of 119 participants in MEBO/PATM cohort).
  Participants from "Non-MEBO Cohort" are not included since they did not participate in the intervention; there was no difference between their entries in terms of flareups or improvements of MEBO/PATM conditions.
Measure: Median (95% Confidence Interval); unit: Normalized OTU counts in gut sample
Units Other Than Participants: samples
Groups:
- MEBO/PATM Subcohort After Flare-up: study participants who experienced flare-ups of MEBO/PATM followed by improvements of their condition documented by corresponding gut samples and QoL questionnaire responses (22 out of 119 in MEBO/PATM cohort)
- MEBO/PATM Subcohort After Improvement: same study participants who experienced improvement in MEBO/PATM status after flare-ups of this condition and submitted corresponding gut samples and QoL questionnaire responses to document their improvement (22 out of 119 in MEBO/PATM cohort)
Arm/Group | MEBO/PATM Subcohort After Flare-up | MEBO/PATM Subcohort After Improvement
Number analyzed (Participants) | 22 | 22
Number analyzed (samples) | 43 | 43
Normalized OTU counts in gut sample
  Selected dermatological bacteria, normalized counts | 162 [135 to 502] | 15 [6 to 110]
  Corynebacteriales order, normalized counts | 302 [300 to 1148] | 91 [85 to 172]
Statistical Analysis 1: Comparison: MEBO/PATM Subcohort After Flare-up vs MEBO/PATM Subcohort After Improvement; Test type: Superiority — Paired Wilcoxon Signed-Rank Tests; p = 0.02, Wilcoxon (Mann-Whitney) — Original p-value for dermatological bacteria was 6e-05. It was adjusted first by applying centered log-ratio (CLR) transformation approach then by false discovery rate (FDR) correction for multiple comparisons by using Benjamini-Hochberg Procedure; Median Difference (Final Values) = 79, 95% CI 2-sided [26 to 163]

5. Secondary Outcome: Alpha Diversity
Description: Alpha (within-sample) diversity measure using microbial abundance information in a phylogenetic framework. Represented by abundance-weighted phylogenetic entropy.
Time Frame: 1 year
Population: Participants that submitted valid stool samples. Since 16 individuals who observed improvement of their symptoms changed the status of their MEBO/PATM condition from "active" to "remission/regression", their samples were grouped in two subgroups (38+33+23+6 = 84+16) Units analyzed represents samples submitted, 233 total.
Measure: Mean (95% Confidence Interval); unit: unitless
Units Other Than Participants: gut microbiome samples
Groups:
- Subjects With Active MEBO: Individuals experiencing uncontrollable episodes of malodor that did not self-diagnose PATM
- Subjects With Active PATM: Individuals experiencing uncontrollable episodes of PATM with or without malodor
- Subjects in Regression or Remission: Individuals self-reporting remission or regression of MEBO/PATM (lessening of the severity or disappearance of the symptoms)
- Non MEBO/PATM Cohort: individuals that never experienced MEBO/PATM episodes
Arm/Group | Subjects With Active MEBO | Subjects With Active PATM | Subjects in Regression or Remission | Non MEBO/PATM Cohort
Number analyzed (Participants) | 38 | 33 | 23 | 6
Number analyzed (gut microbiome samples) | 97 | 85 | 35 | 16
unitless | 1.7 [1.6 to 1.8] | 1.6 [1.0 to 2.2] | 1.7 [1.6 to 1.8] | 1.9 [1.8 to 2.0]

ADVERSE EVENTS:
Time Frame: participants were observed for one year
Groups:
- Study Participants: The cohort is individuals who consented to submit stool samples, including those who experienced symptoms of idiopathic malodor or PATM ("people allergic to me" condition) and received the support-group intervention.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT03582826/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03582826/ICF_001.pdf